CLINICAL TRIAL: NCT03020979
Title: A Phase II, Single-Arm, Open-Label, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Apatinib in Patients With Refractory Malignant Ascites
Brief Title: A Clinical Trial With Apatinib for Subjects With Refractory Malignant Ascites
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Qiong Wu, M.D. Ph.D., The First Affiliated Hospital of Bengbu Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BYEC20161201
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Malignant Ascites; Apatinib
MeSH Terms: interventions — apatinib

ARMS (1):
- 500mg apatinib (Experimental): Patients will receive 500mg of apatinib tablet orally, once daily.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Patients will take 500mg apatinib daily orally.

SUMMARY:
Malignant ascites is a severe complication of many types of human cancer. Animal and clinical analyses have shown that angiogenesis plays a critical role in the formation of malignant ascites. Therefore, drugs such as apatinib that target angiogenesis may control the development of malignant ascites. The study is to evaluate the efficacy and safety of apatinib in patients with refractory malignant ascites.

DETAILED DESCRIPTION:
The study is to investigate the efficacy and safety of apatinib in patients with refractory malignant ascites. A total of 120 patients with performance status 0-2 were enrolled in this study and 500mg apatinib tablets were administered orally, once daily until disease progression or intolerable toxicity or patients withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or symptomatic ascites with positive cytology secondary to any histologically confirmed tumor type not amenable to cytoreductive surgery or additional chemotherapy
* Patients may enroll in this study irrespective of previous therapy including diuretics, surgery, chemotherapy, immunotherapy and radiation therapy
* Must have received a minimum of two paracentesis procedures and a trial of diuretic therapy within 60 days of study entry
* Age Restrictions: 18-75 years
* Life Expectancy: 12 weeks or more
* ECOG Performance Status: 0-2
* Able and willing to provide informed consent and comply with study and/or follow-up procedures
* Normal organ and marrow function as defined by: Leukocytes >/= 3,000/mcL; Absolute neutrophil count >/= 1,500/mcL; Platelets >/= 100,000/mcL; Total bilirubin within normal institutional limits; AST (SGOT)/ALT(SGPT) </= 2.5 X institutional upper limit of normal (ULN); Creatinine within normal institutional limits OR Creatinine clearance >/+ 60 mL/min for patients with creatinine levels above the institutional normal; Serum Potassium within normal institutional limits; Serum Sodium within normal institutional limits

Exclusion Criteria:

* Patients having received anti-angiogenic agents as part of the treatment of their malignancy within 60 days prior to study entry
* Current, recent (within 30 days of the first infusion of this study) or planned administration of chemotherapy (including all routes of administration), immunotherapy, biologic therapy, radiation therapy or any other anti-angiogenic therapy (e.g., bevacizumab, other tyrosine kinase inhibitors)
* Current, recent (within 30 days of the first infusion of this study), or planned participation in any other experimental drug study
* Pregnant women; A serum pregnancy test will be given to females of childbearing potential prior to study enrollment and the participant must agree to use adequate contraception (barrier or hormonal methods) prior to study entry and for the duration of study participation.
* Un-controlled hypertension (defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg
* History of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade III or greater congestive heart failure
* History of myocardial infarction, unstable angina, stroke or transient ischemic attack within 6 months prior to study entry
* Known CNS disease, except for treated brain metastasis.
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study entry
* History of gastrointestinal hemorrhage within 6 month prior to study entry
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study entry or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device or paracentesis/thoracentesis, within 7 days prior to study entry
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to study entry
* Any bowel obstruction that has not fully recovered despite medical or surgical intervention prior to study entry
* Evidence of bowel wall thickening outside the site of the known primary malignancy on baseline radiographs
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a Urine Protein/Creatinine ration >/= 1.0 at screening
* Known hypersensitivity to any component of apatinib.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The repeat paracentesis response rate (proportion of subjects who have a doubling of baseline time to repeat paracentesis) | 12 weeks after initiation of study treatment

SECONDARY OUTCOMES:
The time to the need for the first repeat abdominal paracentesis after the start of apatinib therapy as compared with historical control data. | 12 weeks after initiation of study treatment
The mean number of paracentesis procedures required in each patient over the course of three months. | 12 weeks after the initiation of study treatment
The effect of apatinib therapy on quality of life in patients with malignant ascites by using EORTC QLQ-C30 V3.0. | 12 weeks after the initiation of study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Qiong Wu, Bengbu, Anhui, China